CLINICAL TRIAL: NCT03008174
Title: Early Speech With One-Way Speaking Valve in Tracheostomy Patients - Pilot Study
Brief Title: Early Speech With One-Way Speaking Valve in Tracheostomy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00080981
Record Dates: First submitted 2016-11-28; First posted 2017-01-02 (Estimated); Results first posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Respiratory Failure; Speech; Aphonia
Keywords: tracheostomy; quality of life; speaking valve; speech; mechanically ventilated patients
MeSH Terms: conditions — Respiratory Insufficiency; Speech; Aphonia | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): 1. Early one-way speaking valve (OWSV) assessment by speech language pathologist (SLP) following 12-24 hours after percutaneous tracheostomy procedure.
  2. Second OWSV evaluation with SLP following 48-60 hours from initial percutaneous tracheostomy procedure.
  3. Third OWSV evaluation with SLP following first tracheostomy tube change. Participants may receive additional SLP sessions between second and third sessions per standard of care.
  Interventions: Other: Early one-way speaking valve (OWSV) assessment
- Control (No Intervention): 1. Standard OWSV evaluation with SLP following 48-60 hours from initial percutaneous tracheostomy procedure.
  2. Second OWSV evaluation with SLP following first tracheostomy tube change. Participants may receive additional SLP sessions between first and second sessions per standard of care.

INTERVENTIONS:
Other: Early one-way speaking valve (OWSV) assessment — The OWSV assessment by speech language pathologists will be completed at 12-24 hours following percutaneous tracheostomy procedure, which is earlier than the current standard of care of 48 hours or later.
  Arms: Intervention

SUMMARY:
Patients with tracheostomy who are on and off of mechanical ventilation initially lose the ability to speak, and the use of one-way speaking valves (OWSV) is one method of restoring speech in these patients. Patients with tracheostomy who experience loss of speech report frustration and feelings of confinement from patients' communication impairment, therefore investigators would like to restore speech in these patients as soon as it is safe to do so. However, there is currently little known in the literature about the timing of the use of OWSV in patients with tracheostomy. Therefore, the investigators propose a pre-test post-test clinical trial pilot study to investigate the safety of early use of OWSV in patients undergoing a percutaneous tracheostomy. Study aims are to identify patients who would benefit from the early use of OWSV and to determine the effects of early use of OWSV on speech and clinical outcomes. To achieve these aims, patients who undergo percutaneous tracheostomy will be screened, and patients meeting screening criteria will be randomized into intervention and control groups. The intervention group will receive early speech-language pathology (SLP) evaluation and OWSV trial at 12-24 hours following tracheostomy procedure, and the control group will receive standard SLP evaluation and OWSV trial at 48-60 hours following tracheostomy procedure. Intervention and control groups will been compared on speech and clinical outcomes measures from pre-test at 12-24 hours following tracheostomy and post-test at 48-60 hours following tracheostomy and characteristics of patients who successfully tolerate early OWSV use will be identified.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received a percutaneous tracheostomy
* Glasgow Coma Scale score ≥9
* Confusion Assessment Method -ICU (CAM-ICU): negative
* Richmond Agitation Sedation Scale (RASS): -1 to +1
* Able to understand English

Exclusion Criteria:

* Open tracheostomy
* Laryngectomy
* Presently using OWSV or capped trach
* Foam-filled cuffed tracheostomy tube
* Presence of known severe airway obstruction
* Presence of post-operative bleeding requiring transfusion or packing
* Presence of air-leak around the cuff resulting in respiratory decompensation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2019-11-28 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinciya Pandian, PhD, MSN, ACNP, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
Will not be sharing data

REFERENCES:
- [Background] Hess DR, Altobelli NP. Tracheostomy tubes. Respir Care. 2014 Jun;59(6):956-71; discussion 971-3. doi: 10.4187/respcare.02920. PMID 24891201
- [Background] Mehta AB, Syeda SN, Bajpayee L, Cooke CR, Walkey AJ, Wiener RS. Trends in Tracheostomy for Mechanically Ventilated Patients in the United States, 1993-2012. Am J Respir Crit Care Med. 2015 Aug 15;192(4):446-54. doi: 10.1164/rccm.201502-0239OC. PMID 25955332
- [Background] Carroll SM. Silent, slow lifeworld: the communication experience of nonvocal ventilated patients. Qual Health Res. 2007 Nov;17(9):1165-77. doi: 10.1177/1049732307307334. PMID 17968034
- [Background] Foster A. More than nothing: the lived experience of tracheostomy while acutely ill. Intensive Crit Care Nurs. 2010 Feb;26(1):33-43. doi: 10.1016/j.iccn.2009.09.004. Epub 2009 Nov 11. PMID 19910195
- [Background] Freeman BD, Isabella K, Lin N, Buchman TG. A meta-analysis of prospective trials comparing percutaneous and surgical tracheostomy in critically ill patients. Chest. 2000 Nov;118(5):1412-8. doi: 10.1378/chest.118.5.1412. PMID 11083694
- [Background] Pandian V, Thompson CB, Feller-Kopman DJ, Mirski MA. Development and validation of a quality-of-life questionnaire for mechanically ventilated ICU patients. Crit Care Med. 2015 Jan;43(1):142-8. doi: 10.1097/CCM.0000000000000552. PMID 25072754
- [Derived] Martin KA, Cole TDK, Percha CM, Asanuma N, Mattare K, Hager DN, Brenner MJ, Pandian V. Standard versus Accelerated Speaking Valve Placement after Percutaneous Tracheostomy: A Randomized Controlled Feasibility Study. Ann Am Thorac Soc. 2021 Oct;18(10):1693-1701. doi: 10.1513/AnnalsATS.202010-1282OC. PMID 33760713

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: 1. Early one-way speaking valve (OWSV) assessment by speech language pathologist (SLP) following 12-24 hours after percutaneous tracheostomy procedure.
  2. Second OWSV evaluation with SLP following 48-60 hours from initial percutaneous tracheostomy procedure.
  3. Third OWSV evaluation with SLP following first tracheostomy tube change. Participants may receive additional SLP sessions between second and third sessions per standard of care.
  Early one-way speaking valve (OWSV) assessment: The OWSV assessment by speech language pathologists will be completed at 12-24 hours following percutaneous tracheostomy procedure, which is earlier than the current standard of care of 48 hours or later.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 10 | 10
Completed | 7 | 6
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (19.7) | 50.6 (16.1) | 50.35 (17.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 4 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3 | 6 | 9
  Caucasian | 6 | 3 | 9
  Hispanic | 0 | 1 | 1
  Middle Eastern | 1 | 0 | 1
Sequential Organ Failure Assessment (SOFA) Score [Mean (Standard Deviation); unit: score on a scale] — The Sequential Organ Failure Assessment (SOFA) score is a scoring system that assesses the performance of several organ systems in the body (neurologic, blood, liver, kidney, and blood pressure/hemodynamics) and assigns a score based on the data obtained in each category. SOFA scores will be reported on a scale of 0 - 24. The lower the score, the patient is not sick and the higher the score, the patient is sicker.
  score on a scale | 5.6 (2.17) | 6.0 (1.63) | 5.8 (1.88)

OUTCOME MEASURES:

1. Primary Outcome: Speech Intelligibility as Assessed by Speech Intelligibility Test Score
Description: Speech intelligibility test scores will be reported in percentages (Percentage of words that were intelligible).
Time Frame: Up to 24 hours after percutaneous tracheostomy procedure (assessed once within the period)
Measure: Mean (Standard Deviation); unit: Percentage of intelligible words
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
Percentage of intelligible words | 25.71 (33.35) | 0 (0)

2. Primary Outcome: Speech Intelligibility as Assessed by Speech Intelligibility Test Score
Description: Speech intelligibility test scores will be reported in percentages (Percentage of words that were intelligible).
Time Frame: Between 25 and 60 hours after percutaneous tracheostomy procedure (assessed once within the period)
Measure: Mean (Standard Deviation); unit: Percentage of intelligible words
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
Percentage of intelligible words | 13 (26.46) | 33.63 (33.12)

3. Primary Outcome: Speech Intelligibility as Assessed by Speech Intelligibility Test Score
Description: Speech intelligibility test scores will be reported in percentages (Percentage of words that were intelligible).
Time Frame: Between 61 hours and 21 days after percutaneous tracheostomy procedure (assessed once within the period)
Population: Data for this outcome measure was only obtained from participants that completed the study.
Measure: Mean (Standard Deviation); unit: Percentage of intelligible words
Arm/Group | Intervention | Control
Number analyzed (Participants) | 7 | 6
Percentage of intelligible words | 74.54 (21.03) | 35.97 (39.5)

4. Secondary Outcome: Quality of Life as Assessed by Quality of Life in Mechanically Ventilated Patients Scores
Description: Quality of life as assessed by Quality of Life in Mechanically Ventilated Patients Scores. QOL scores will be reported on a scale of 0 - 100. The lower the score, the poorer the quality of life is, and the higher the score, the better the quality of life.
Time Frame: Up to 24 hours after percutaneous tracheostomy procedure (assessed once within the period)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
score on a scale | 42.0 (18.0) | 41.7 (13.4)

5. Secondary Outcome: Quality of Life as Assessed by Quality of Life in Mechanically Ventilated Patients Scores
Description: as for outcome 4
Time Frame: Between 25 and 60 hours after percutaneous tracheostomy procedure (assessed once within the period)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
score on a scale | 53.1 (24.8) | 47.3 (12.8)

6. Secondary Outcome: Quality of Life as Assessed by Quality of Life in Mechanically Ventilated Patients Scores
Description: as for outcome 4
Time Frame: Between 61 hours and 21 days after percutaneous tracheostomy procedure (assessed once within the period)
Population: Data for this outcome measure was only obtained from participants that completed the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention | Control
Number analyzed (Participants) | 7 | 6
score on a scale | 55.0 (22.0) | 47.1 (16.2)

7. Secondary Outcome: Number of Participants With Bleeding
Description: Bleeding will be reported as present or absent.
Time Frame: At the time of use of speaking valve up to 24hours after percutaneous tracheostomy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Bleeding
Description: Bleeding will be reported as present or absent.
Time Frame: At the time of use of speaking valve between 25 and 60 hours after percutaneous tracheostomy procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Bleeding
Description: Bleeding will be reported as present or absent.
Time Frame: At the time of use of speaking valve between 61 hours and 21 days after percutaneous tracheostomy procedure
Population: Data for this outcome measure was only obtained from participants that completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

10. Secondary Outcome: Intensive Care Unit (ICU) Length of Stay
Description: ICU length of stay will be reported in days.
Time Frame: At the time of discharge, up to 4 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
Days | 51 (30.37) | 53.9 (51.46)

11. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay will be reported in days.
Time Frame: At the time of discharge, up to 4 months
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 10 | 10
Days | 69.7 (33.86) | 75.6 (101.12)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT03008174/Prot_SAP_000.pdf